CLINICAL TRIAL: NCT06539364
Title: The Effect Of Surgical And Non-Surgical Periodontal Treatment On The Quality Of Life In Patients With Periodontitis.
Brief Title: Effects Of Different Periodontal Treatments On Quality Of Life In Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Aliye Gerzile, Research Assistant, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-gokae-1095
Record Dates: First submitted 2024-07-17; First posted 2024-08-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Quality of Life
Keywords: periodontitis; quality of life; VAS; OHIP-14; OHRQoL-UK
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: According to full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL),bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were obtained from 50 systemically healthy individuals with periodontitis and after the initial treatment repeat measurements were taken at the control session to evaluate participation in the surgical treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NON-SURGICAL PERIODONTAL TREATMENT (Active Comparator): Patients included in this group underwent full-mouth scaling followed by root planning in the necessary areas. At the 3-week follow-up session, periodontal surgery was not planned. Periodontal records were maintained, and surveys were administered at follow-up visits.
  Interventions: Diagnostic Test: Quality of life surveys were conducted
- SURGICAL PERIODONTAL TREATMENT (Experimental): Patients included in this group received full-mouth scaling followed by root planning in the necessary areas. After a 3-week follow-up period, periodontal records were taken and surgical periodontal treatment was administered to the required areas. Periodontal records were maintained and surveys were conducted at follow-up visits.
  Interventions: Diagnostic Test: Quality of life surveys were conducted

INTERVENTIONS:
Diagnostic Test: Quality of life surveys were conducted — Quality of life surveys were conducted with OHIP-14, OHRQoL-UK and VAS

SUMMARY:
In this study, the quality of life of patients with stage 3 grade C periodontitis who underwent surgical and non-surgical periodontal treatments was evaluated. Patients were compared based on their quality of life using OHIP-14 and OHRQoL-UK questionnaires, as well as a VAS scale, against those who did not receive periodontal treatment, those who received only phase 1 treatment one month prior, and those who underwent periodontal surgical treatment three months prior.

DETAILED DESCRIPTION:
Currently, the most commonly used reliable scales to measure oral health-related quality of life are the OHIP-14 (Oral Health Impact Profile) and OHRQoL-UK questionnaires. Fifty patients with stage 3 and grade c whose clinical periodontal records (PI, GI, PD and BOP) were obtained were included in the study. OHRQoL-UK, OHIP-14 questionnaires and VAS were applied at the first session (T1). Initial periodontal treatment (scaling, polishing and oral hygiene education) was performed, and non-surgical periodontal treatment (root surface debridement under local anesthesia) was performed in the next session. Three to four weeks after this treatment, patients were recalled for follow-up and all clinical indices and questionnaires were repeated (T2). After re-evaluation, the patients were divided into a surgical group (23 patients) and a non-surgical group (27 patients). Open flap debridement was performed in areas requiring surgery (radiologic bone loss and SCD>5mm). Patients were recalled 12-14 weeks after surgery and all indices and questionnaires were repeated (T3).

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Over 18 years of age
* Willing to voluntarily participate in the study
* No mental retardation or any other disorder that would impede communication

Exclusion Criteria:

* Presence of any systemic disease affecting periodontal tissues or use of medication that impacts periodontal health
* Pregnancy or lactation
* Having undergone periodontal treatment in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
obtain survey results | Baseline (T1), 3 weeks after non-surgical periodontal treatment (T2), and 12 weeks after surgical periodontal treatment (T3).
  obtaining survey results to see the impact on patients' quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Gerzile A, Naziker Y, Ozer E, Ertugrul AS. Impact of Surgical and Non-Surgical Periodontal Therapy on Quality of Life in Case of Periodontitis. Oral Dis. 2025 Aug;31(8):2564-2571. doi: 10.1111/odi.15316. Epub 2025 Mar 19. PMID 40106822